CLINICAL TRIAL: NCT02365480
Title: Phase I Trial of Berberine in Subjects With Ulcerative Colitis
Brief Title: Berberine Chloride in Preventing Colorectal Cancer in Patients With Ulcerative Colitis in Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2015-00173; NCI-2015-00173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2014-03-01 (Other: Northwestern University); NWU2014-03-01 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-19 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (berberine chloride) (Experimental): Patients receive berberine chloride PO TID for 90 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berberine Chloride; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Participants receive placebo PO TID for 90 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Drug: Berberine Chloride — Given PO
  Other Names: Berberine Chloride Dihydrate; Berberine Hydrochloride; Berberinum Chloride
  Arms: Arm I (berberine chloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)

SUMMARY:
This randomized, pilot phase I trial studies the side effects of berberine chloride in treating patients with ulcerative colitis and who are in remission (a decrease in or disappearance of signs and symptoms of cancer) to reduce the risk of colorectal cancer. Patients with ulcerative colitis are at increased risk for colorectal cancer. Chemoprevention is the use of drugs, such as berberine chloride, to keep a disease/condition from forming or coming back. The use of berberine chloride may keep colorectal cancer from forming in patients with ulcerative colitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of berberine (berberine chloride) administered to participants with ulcerative colitis (UC) in clinical remission while receiving maintenance therapy with mesalamine.

SECONDARY OBJECTIVES:

I. Determine the molecular efficacy of berberine by examining the following biomarkers:

* Plasma-based measures of inflammation, including the blood C-reaction protein (CRP) level, erythrocyte sedimentation rate (ESR), and cytokines such as TNFa, IL-4, IL-6, IL-8 and IL-10 measured by enzyme-linked immunosorbent assay (ELISA).
* Tissue-based measures of inflammation, including TNFα, COX-2, and NF-kappa (κ)B by immunohistochemistry (IHC), and anti-cancer action, including antigen Ki-67 (Ki67) and activated caspase-3 by IHC, and deoxyribonucleic acid (DNA) methylation on SFRP1, TCERG1L FBN2, TFPI2 using the methylation-specific polymerase chain reaction (qMSP) strategy.

II. Clinical efficacy: UC related symptoms will be measured using the Ulcerative Colitis Disease Activity Index (i.e. the Mayo score) (UCDAI).

III. Histological analysis for inflammation: severity of histologic inflammation will be evaluated using the Geboes grading system.

IV. Determine plasma concentration of berberine.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive berberine chloride orally (PO) thrice daily (TID) for 90 days in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive placebo PO TID for 90 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are follow-up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis in clinical remission (UCDAI) =< 1 for at least 3 months, regardless of how long ago they were diagnosed for UC
* Receiving maintenance therapy with mesalamine for at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin within normal institutional limits; higher values (=< 3 x institutional upper limit of normal [ULN]) are acceptable in participants with: 1. known or suspected cholangitis associated with Crohn's disease, or 2, known or suspected inborn errors of metabolism that lead to increased bilirubin
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOP])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional ULN
* Creatinine within normal institutional limits
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had any immunomodulatory treatment in the past 3 months will be excluded
* Participants who have taken any medicines that are inducers, inhibitors or substrates of select cytochrome (CYP) isozymes within the past 3 months will be excluded; participants who have consumed either grapefruit juice or Seville orange juice in the past 7 days will be excluded
* Participants with dysplasia-associated mass or lesion (DALM) due to longstanding idiopathic inflammatory bowel disease will be excluded
* Participants who are currently receiving any other investigational agents or have received investigational agents within the past 3 months will be excluded
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to berberine will be excluded
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that in the opinion of investigators would jeopardize patient safety of data integrity are excluded; individuals who are human immunodeficiency virus (HIV) positive will not necessarily be excluded, will be considered on a case-by-case basis, but will be required to meet criteria related to patient safety and data integrity, as assessed by investigators
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with berberine; women are considered to be of child-bearing potential if they are not surgically sterile or under the age 65 and have menstruated within the last two years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Principal Investigator — Northwestern University
Locations (2):
- Northwestern University, Chicago, Illinois, United States
- Fourth Military Medical University, Xi'an, Shaanxi, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened to accrual 06/16/2016 and closed to accrual 10/18/2017. All participants were recruited at Xijing Hospital, Xi'an, China.
Pre-assignment Details: Twenty participants were screened and eighteen were randomized and began study intervention.
Period: Overall Study
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Started | 14 | 4
Completed | 12 | 4
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 14 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 4 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 14 | 4 | 18
BMI [Median (Inter-Quartile Range); unit: kilogram per square meter] — Body Mass Index
  kilogram per square meter | 23.5 [19.9 to 24.4] | 22.8 [20.3 to 25.1] | 23.5 [19.7 to 24.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Toxicity Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version (v.) 4.0
Description: Relevant counts and rates will be evaluated and reported by standard clinical tests. Symptoms such as fever, fatigue, weight loss, appetite, stool frequency, bloody stool and other upper and lower gastrointestinal tract symptoms in participants will be observed and recorded.
Time Frame: Baseline up to 30 days post-treatment (up to 120 days total)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 14 | 4
Participants | 2 | 0

2. Primary Outcome: Number of Participants With Organ Toxicity Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version (v.) 4.0
Description: Evaluated by standard clinical tests. Symptoms such as fever, fatigue, weight loss, appetite, stool frequency, bloody stool and other upper and lower gastrointestinal tract symptoms in participants will be observed and recorded.
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 14 | 4
Participants | 2 | 0

3. Secondary Outcome: Clinical Efficacy of Berberine Chloride Measured Using the UCDAI Score
Description: UC related symptoms measured using the Ulcerative Colitis Disease Activity Index [UCDAI]. Score results may range from 0 to 12. 0 indicates normal disease and a higher score up to 12 indicates severe disease.
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 4
score on a scale
  Baseline | 0.83 (0.37) | 1 (0)
  Day 90 (end of intervention) | 0.5 (0.5) | 0.5 (0.5)
Statistical Analysis 1: Comparison: Arm I (Berberine Chloride) vs Arm II (Placebo); Test type: Other; p = 0.60, Fisher Exact; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.10 to 36.37]

4. Secondary Outcome: Change in Plasma Markers of Inflammation Via ELISA
Description: TNF-α, a cytokine plasma-based measure of inflammation, measured by enzyme linked immunosorbent assay (ELISA). A numeric value in pg/mL.
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 4
pg/mL
  Baseline | 61.47 (22.47) | 58.68 (22.35)
  Day 90 (end of intervention) | 55.06 (19.20) | 54.68 (3.21)

5. Secondary Outcome: Change in Colorectal Tissue Biomarkers Expression by IHC
Description: Ki-67, a tissue based measure of inflammation, staining was graded and scored on a scale. The higher the score, the greater the expression of Ki-67:
  0 = no cells stained
  1. = 1/3 of cells stained
  2. = 1/2 of cells stained
  3. = ≥ 2/3 of cells stained
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 4
score on a scale
  Baseline | 1.83 (0.90) | 2.25 (0.43)
  Day 90 (end of intervention) | 1.33 (0.47) | 1.5 (0.87)

6. Secondary Outcome: Change in Blood Berberine Chloride Concentration Measurement Using High-performance Liquid Chromatography/Mass Spectrometry
Description: Change in blood berberine chloride concentration measurement measured using high-performance liquid chromatography/mass spectrometry.
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 4
ng/ml
  Baseline | 0.20 (0.21) | 0.09 (0.04)
  Day 90 (end of intervention) | 1.16 (1.28) | 0.18 (0.19)

7. Secondary Outcome: Severity of Histologic Inflammation
Description: Histologic sections will be stained with hematoxylin and eosin and the severity of histologic inflammation will be evaluated using the Geboes scoring system. The Geboes score is taken as the highest category of change among the following: 0.0-0.3, structural change only; 1.0-1.3, chronic inflammation; 2.0-2.3, lamina propria neutrophils; 3.0-3.3, neutrophils in epithelium; 4.0-4.3, crypt destruction; and 5.0-5.4, erosions or ulcers.
Time Frame: Baseline to Day 90 (end of intervention)
Population: Participants with ulcerative colitis in clinical remission and maintained by Mesalamine.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 4
score on a scale
  Baseline | 2.89 (1.41) | 4.68 (0.58)
  Day 90 (end of intervention) | 2.37 (1.66) | 4.45 (0.92)

ADVERSE EVENTS:
Time Frame: 120 days after randomization
Description: Adverse events deemed possibly, probably, or definitely related to the study intervention by study physician are reported.
Arm/Group | Arm I (Berberine Chloride) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/4
Other Adverse Events (participants affected / at risk) | 1/14 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Berberine Chloride) (N=14) | Arm II (Placebo) (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT02365480/Prot_SAP_000.pdf